CLINICAL TRIAL: NCT02417337
Title: Efficacy of Pain Control Following Root Canal Treatment Using Paracetamol Alone and in Combination With Three Different Non-Steroidal Anti-Inflammatory Analgesics
Brief Title: Efficacy of Different Drugs to Control Post Root Canal Treatment Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Khartoum (Other)
Responsible Party: Principal Investigator, Dr. Wail Elzaki, Lecturer at Faculty of Dentistry, University of Khartoum
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: University of Khartoum
Record Dates: First submitted 2015-03-30; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Pain; Postoperative Pain; Irreversible Pulpitis
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Endodontics; Acetaminophen; Ibuprofen; Mefenamic Acid; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group I (Active Comparator): paracetamol 1000mg
  Interventions: Procedure: Root Canal Treatment; Drug: Paracetamol
- Group II (Experimental): ibuprofen 600mg + paracetamol 1000mg,
  Interventions: Procedure: Root Canal Treatment; Drug: Paracetamol; Drug: Ibuprofen
- Group III (Experimental): Mefenamic acid 500mg + Paracetamol 1000mg
  Interventions: Procedure: Root Canal Treatment; Drug: Paracetamol; Drug: Mefenamic acid
- Group IV (Experimental): Diclofenac K 50mg + paracetamol 1000 mg
  Interventions: Procedure: Root Canal Treatment; Drug: Paracetamol; Drug: Diclofenac
- Group V (Placebo Comparator): No medication
  Interventions: Procedure: Root Canal Treatment

INTERVENTIONS:
Procedure: Root Canal Treatment — A standardized endodontic procedures performed.
  Other Names: Endodontic treatment
Drug: Paracetamol
  Arms: Group I; Group II; Group III; Group IV
Drug: Ibuprofen
  Arms: Group II
Drug: Mefenamic acid
  Arms: Group III
Drug: Diclofenac
  Arms: Group IV

SUMMARY:
Root canal therapy will ideally eliminate post-endodontic pain but occasionally analgesics are needed to diminish the pain [1]. Development of pain after completion of root canal treatment may undermine patients' confidence in the procedure and the clinician [2]. Non-steroidal anti-inflammatory drugs are one of the most frequently taken analgesic medications for dental pain. Their popularity attributed to their efficacy in relieving pain and fever and low side effect profile at therapeutic doses [3]. Mono-therapy analgesic has a low effect on dental pain. Improvement was performance by combining analgesics with different mechanisms of action without raising any adverse effects [4], was effective in controlling moderate to severe pain. The combination of a non-steroidal anti-inflammatory drug (NSAID) and paracetamol has shown additive analgesia for treating dental pain in several studies [5,6]. Endodontic treatment with a lower prevalence of postoperative pain is usually the treatment of choice. There have been no controlled dental studies evaluating the additive effects of combining a non-steroidal anti-inflammatory drug with paracetamol. Breivik et al [6] & Menhinick et al [7] found that a combination of acetaminophen and ibuprofen was more effective than ibuprofen alone in managing postoperative pain. Aim of the present study, to evaluate the efficacy of the paracetamol when used alone and in combinations with three groups of drugs to control postoperative endodontic pain.

DETAILED DESCRIPTION:
Background: Management of pain is challenging part of dental treatment, sometimes pain is a major postoperative symptom after many dental procedures especially for endodontics. The aim of the present randomized clinical trial was to investigate the efficacy of using paracetamol alone and three combinations of non-steroidal anti-inflammatory drugs with paracetamol, to control postoperative endodontics pain.

Methodology: 185 patients who had anterior or premolar teeth with irreversible pulpitis without any signs and symptoms of apical periodontitis and with moderate to severe pain. Patients were divided by allocation randomization into five groups. Four experimental groups receiving different medication; group I (single dose of paracetamol); group II (ibuprofen / paracetamol); group III (diclofenac k / paracetamol), group IV (mefenamic acid /paracetamol) and group V (no medication group). The groups received the medication after the first appointment where the pulp removed, and canals fully prepared. Pain intensity was scored based on 10-point VAS before and after treatment for up to 8 hours postoperatively. Sign test used for comparing pain score before and after treatment. This randomized control clinical trial was conducted on patients who were considered potential candidates if they had moderate to severe spontaneous pain of odontogenic origin (40-100 mm on a visual analogue scale, VAS). Patients were selected from those attending the Conservative dentistry clinics in both the University and the Teaching Hospital Emergency Clinic.

The medications were prepared in the laboratories of faculty of Pharmacy. Four groups of medications were prepared as follows; Group I: paracetamol 1000mg Group II: ibuprofen 600mg + paracetamol 1000mg, Group III: Mefenamic acid 500mg + Paracetamol 1000mg Group IV: Diclofenac K 50mg + paracetamol 1000 mg

ELIGIBILITY:
Inclusion Criteria:

1. Patient reported spontaneous pain moderate to severe, ranging from 50 to 100 mm on a VAS (0-100 mm);
2. Adult patients presented for emergency endodontic treatment with a symptomatic maxillary or mandibular tooth (anterior and premolar) with a pulpal diagnosis of Irreversible pulpitis and normal periapex.
3. Patient choose to have root canal treatment for pain of endodontic origin.
4. The patient presented with American Society of Anesthesiologists (ASA) I or II medical history (ASA 1963).
5. The patient had read and thoroughly understood the pain score level sheet

Exclusion Criteria:

1. Patients below 18 years of age;
2. Analgesic taken within the last 4 hours;
3. History of allergy to NSAIDs, paracetamol or local anaesthetics;
4. History of uncontrolled systemic disease [gastrointestinal (GI) disorders, oesophageal reflux, active asthma, decreased hepatic function, haemorrhagic disorders, or poorly controlled diabetes mellitus].
5. Patients currently taking opioids, monoamine oxidase inhibitors, tricyclic antidepresssants, carbamazepine, diuretics, or anticoagulants;
6. There was history of opioid addiction or abuse; and
7. Pregnant or nursing female patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of different Drugs to Control Post Root Canal Treatment Pain as measured by Visual Analogue Scale. | 8 hours
  The patients were asked to make entries on the VAS (numerical score) every hour for the first 4 hours after taking the medication and then every 2 hours following that; a total of six entries over 8 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Khartoum, Faculty of Dentistry,, Khartoum, Khartoum State, Sudan

REFERENCES:
- [Result] Owatz CB, Khan AA, Schindler WG, Schwartz SA, Keiser K, Hargreaves KM. The incidence of mechanical allodynia in patients with irreversible pulpitis. J Endod. 2007 May;33(5):552-6. doi: 10.1016/j.joen.2007.01.023. Epub 2007 Mar 6. PMID 17437870
- [Result] Albashaireh ZS, Alnegrish AS. Postobturation pain after single- and multiple-visit endodontic therapy. A prospective study. J Dent. 1998 Mar;26(3):227-32. doi: 10.1016/s0300-5712(97)00006-7. PMID 9594474
- [Result] Attar S, Bowles WR, Baisden MK, Hodges JS, McClanahan SB. Evaluation of pretreatment analgesia and endodontic treatment for postoperative endodontic pain. J Endod. 2008 Jun;34(6):652-5. doi: 10.1016/j.joen.2008.02.017. Epub 2008 Apr 2. PMID 18498882
- [Result] Mehlisch DR. The efficacy of combination analgesic therapy in relieving dental pain. J Am Dent Assoc. 2002 Jul;133(7):861-71. doi: 10.14219/jada.archive.2002.0300. PMID 12148679
- [Result] Breivik EK, Barkvoll P, Skovlund E. Combining diclofenac with acetaminophen or acetaminophen-codeine after oral surgery: a randomized, double-blind single-dose study. Clin Pharmacol Ther. 1999 Dec;66(6):625-35. doi: 10.1053/cp.1999.v66.103629001. PMID 10613619
- [Result] Keiser K, Hargreaves K.Building effective strategies for the management of endodontic pain. Endodontic Topics, Volume 3, Issue 1, pages 93-105, November 2002
- [Result] Menhinick KA, Gutmann JL, Regan JD, Taylor SE, Buschang PH. The efficacy of pain control following nonsurgical root canal treatment using ibuprofen or a combination of ibuprofen and acetaminophen in a randomized, double-blind, placebo-controlled study. Int Endod J. 2004 Aug;37(8):531-41. doi: 10.1111/j.1365-2591.2004.00836.x. PMID 15230906
- [Derived] Elzaki WM, Abubakr NH, Ziada HM, Ibrahim YE. Double-blind Randomized Placebo-controlled Clinical Trial of Efficiency of Nonsteroidal Anti-inflammatory Drugs in the Control of Post-endodontic Pain. J Endod. 2016 Jun;42(6):835-42. doi: 10.1016/j.joen.2016.02.014. Epub 2016 Apr 12. PMID 27080115